CLINICAL TRIAL: NCT01510509
Title: TITANIC-XV Trial: Prospective, Multicenter and Randomized Trial (Bioactive Bare Metal Titanium Stent Versus Everolimus Drug Eluting Stent)
Brief Title: The Titan Versus Everolimus Intracoronary Stent (Xience V) in Diabetic Patients
Acronym: TITANIC-XV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario Infanta Cristina (Other)
Responsible Party: Principal Investigator, Jose Ramon Lopez Minguez, MD, PhD, Chief of Interventional Cardiology Deparment, Hospital Universitario Infanta Cristina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TITANIC-XV
Record Dates: First submitted 2012-01-11; First posted 2012-01-16 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2008-12

CONDITIONS: Diabetes Mellitus; Percutaneous Coronary Intervention
Keywords: Drug Eluting Stent; Bioactive Bare Metal Stent
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Titanium bare metal stent (Experimental): Titanium bare metal stent (Titan2®, Hexacath, Paris, France)
  Interventions: Device: Titanium bare metal stent (Titan2®)
- Everolimus Drug Eluting Stent (Experimental): Xience-V®, Abbott Vascular, Santa Clara, California, USA
  Interventions: Device: Everolimus Drug Eluting Stent (Xience-V®)

INTERVENTIONS:
Device: Titanium bare metal stent (Titan2®) — Titan2®, Hexacath, Paris, France
  Arms: Titanium bare metal stent
Device: Everolimus Drug Eluting Stent (Xience-V®) — Xience-V®, Abbott Vascular, Santa Clara, California, USA
  Arms: Everolimus Drug Eluting Stent

SUMMARY:
Even though the safety of drug eluting stents has been long established, in roughly 25% o patients their implantation is not considered, for specifically clinical reasons (chronic anticoagulation, bleeding, etc…), which make prolonged use of clopidogrel unsuitable. A considerable percentage of these patients have diabetes mellitus, a well known risk factor for stent thrombosis. Recently, the special characteristics of the titanium stent with nitric oxide have been described, causing it to be considered as a bioactive stent.

The TITANIC-XV trial was a prospective randomized multi-center active-treatment-controlled clinical trial, with the chief aim to evaluate clinical outcome after titanium bare metal stent (Titan2®, Hexacath, Paris, France) implantation as compared with everolimus drug eluting stent (Xience-V®, Abbott Vascular, Santa Clara, California, USA) in diabetic patients undergoing percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Diabetes mellitus according to the World Health Organization Report
* Percutaneous coronary intervention due to at least one significant de novo lesion (defined as at least 50% diameter stenosis by visual estimation) in a native coronary artery or coronary bypass graft.
* Informed Consent "signed"

Exclusion Criteria:

* Inclusion in another clinical research protocol
* Pregnancy
* STEMI within 48 hours
* Unprotected left main disease
* Restenotic lesions
* Stent diameter < 2,5 mm or > 3,5 mm
* Stent length more than 28 mm in < 3 mm vessels
* Chronic total occlusions
* Allergy to aspirin, clopidogrel, heparin or abciximab
* Active bleeding or a significant increase in bleeding risk
* Significant renal insufficiency defined as creatinine > 2 mg/dl
* Severely depressed LV function (EF≤35%)
* Cardiogenic shock
* Ischemic stroke within the last 6 months
* Contraindication for DES
* Disease with life expectancy < 12 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-01

PRIMARY OUTCOMES:
Major adverse cardiac events
  Comparison of major adverse cardiac events defined as death, non fatal myocardial infarction, brain stroke or new revascularization at 1, 6, 12 and 24 months follow-up between the two treatment strategies.

SECONDARY OUTCOMES:
Late luminal loss
  Comparison of late luminal loss within the in-segment zone at 9 months between the two treatment strategies in the subgroup of patients with angiographic follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Ramon Lopez-Minguez, MD, Principal Investigator — Hospital Universitario Infanta Cristina (Badajoz, Spain). Interventional Cardiology Department.
Locations (8):
- Heart Center, Satakunta Hospital, Pori, Finland, Satakunta, Pori, Finland
- Spain (7):
  - Hospital de Torrevieja, Torrevieja, Alicante
  - Hospital Universitario Infanta Cristina, Badajoz, Badajoz
  - Hospital Puerto Real de Cádiz, Puerto Real, Cadiz
  - Hospital Juan Ramón Jiménez de Huelva, Huelva, Huelva
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Virgen de la Salud de Toledo, Toledo, Toledo
  - Hospital General Universitario de Valencia, Valencia, Valencia